CLINICAL TRIAL: NCT02842242
Title: A Phase 2 Open-label Pilot Study to Evaluate Efficacy, Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of MYK-461 in Subjects With Symptomatic Hypertrophic Cardiomyopathy and Left Ventricular Outflow Tract Obstruction
Brief Title: A Phase 2 Open-label Pilot Study Evaluating MYK-461 in Subjects With Symptomatic Hypertrophic Cardiomyopathy and Left Ventricular Outflow Tract Obstruction
Acronym: PIONEER-HCM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MyoKardia, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MYK-461-004
Record Dates: First submitted 2016-07-20; First posted 2016-07-22 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Cardiomyopathy, Hypertrophic Obstructive; Left Ventricular Outflow Tract Obstruction
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Ventricular Outflow Obstruction, Left | interventions — MYK-461

ARMS (1):
- Open Label (Experimental): MYK-461
  Interventions: Drug: MYK-461

INTERVENTIONS:
Drug: MYK-461

SUMMARY:
The purpose of this phase 2 open-label pilot study is to evaluate the efficacy, pharmacokinetics (PK), pharmacodynamics (PD), safety, and tolerability of MYK-461 in subjects with symptomatic HCM and LVOT obstruction aged 18-70 years.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosed with HCM (hypertrophied and non-dilated left ventricle in absence of systemic or other known cause), with LV wall thickness ≥ 15 mm at time of initial diagnosis or ≥ 13 mm with a positive family history of HCM.
* Age 18-70
* BMI 18-37kg/m2
* Documented LVEF ≥ 55% at the Screening visit as determined by the investigator and the investigational site's echocardiography laboratory.
* Resting LVOT gradient ≥ 30 mg Hg and post-exercise peak LVOT gradient ≥ 50 mm Hg
* NYHA functional class II or higher

Key Exclusion Criteria:

* History of sustained ventricular tachyarrhythmia.
* History of syncope with exercise within past 6 months.
* Active infection.
* Persistent atrial fibrillation or atrial fibrillation at Screening or history of paroxysmal atrial fibrillation with resting rate document > 100bpm within 1 year of screening.
* Has QTc Fridericia (QTcF) > 500 ms, or any other ECG abnormality considered by the investigator to pose a risk to subject safety (e.g. second degree atrioventricular block type II).
* Aortic stenosis or fixed subaortic obstruction.
* History of LV systolic dysfunction (LVEF < 45%) at any time during their clinical course.
* History of obstructive coronary artery disease.
* History or evidence of any other clinically significant disorder, condition, or disease that, in the opinion of the investigator or MyoKardia physician, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion.
* Part A: Ongoing therapy with beta blockers, calcium channel blockers, or disopyramide. Subjects on any of these medications who, in the opinion of the investigator, can safely be withdrawn are eligible as long as medication is discontinued at least 14 days prior to the Screening visit.
* Part B: Ongoing therapy with calcium channel blockers or disopyramide. Subjects on any of these medications who, in the opinion of the investigator, can safely be withdrawn are eligible as long as medication is discontinued at least 14 days prior to the Screening visit.
* Prior treatment with cardiotoxic agents such as doxorubicin or similar, or current treatment with antiarrhythmic drugs that have negative inotropic activity, e.g. flecainide or propafenone.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Sehnert, MD, Study Chair — MyoKardia, Inc.
Locations (7):
- United States (7):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Yale New Haven Hospital, New Haven, Connecticut
  - Tufts Medical Center, Boston, Massachusetts
  - Washington University St. Louis, St Louis, Missouri
  - Duke Health Center at Southpoint, Durham, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Hospital of the University of Pennsylvania (Penn Heart and Vascular Center), Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Heitner SB, Jacoby D, Lester SJ, Owens A, Wang A, Zhang D, Lambing J, Lee J, Semigran M, Sehnert AJ. Mavacamten Treatment for Obstructive Hypertrophic Cardiomyopathy: A Clinical Trial. Ann Intern Med. 2019 Jun 4;170(11):741-748. doi: 10.7326/M18-3016. Epub 2019 Apr 30. PMID 31035291

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: Mavacamten 10 to 20 mg/d without background medications
- Cohort B: Mavacamten 2 to 5 mg/d with beta-blockers allowed.
Period: Overall Study
Arm/Group | Cohort A | Cohort B
Started | 11 | 10
Completed | 10 | 10
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Customized [Mean (Full Range); unit: years]
  Mean Age (range) | 56 [22 to 70] | 58 [26 to 67] | 57 [22 to 70]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 7 | 5 | 12
  Female | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 10 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 11 | 9 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Postexercise LVOT gradient [Mean (Standard Deviation); unit: mm Hg] — Population: Based on available data
  mm Hg
    number analyzed (Participants) | 9 | 9 | 18
    (all) | 103 (50) | 86 (43) | 94.5 (0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Post-exercise Peak LVOT Gradient From Baseline to Week 12
Description: Post-exercise peak LVOT gradients are assessed after a treadmill stress test by echocardiography.
Time Frame: Baseline and Week 12
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 8 | 9
mm Hg | -89.5 [-138.3 to -40.7] | -25.0 [-47.1 to -3.0]

2. Secondary Outcome: Number of Participants Achieving a Post-exercise Peak LVOT Gradient Response of < 30 mmHg. Gradient < 30 mmHg
Description: LVOT gradients are assessed after a treadmill stress test by echocardiography.
Time Frame: Baseline and Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 11 | 10
Participants | 8 | 0

3. Secondary Outcome: Change in Dyspnea Symptom Score From Baseline to Week 12
Description: The scale name is Dyspnea Numeric Rating Scale (NRS). It is intended to measure how much shortness of breath you have had in the past week. 0 = no shortness of breath and 10 = shortness of breath as the worst possible.
Time Frame: Baseline and Week 12
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 10 | 10
units on a scale | -3.1 [-4.1 to -2.1] | -3.0 [-5.0 to -1.0]

4. Secondary Outcome: Change in Peak VO2 From Baseline to Week 12
Description: Peak VO2 is assessed using a cardiopulmonary exercise test.
Time Frame: Baseline and Week 12
Measure: Mean (95% Confidence Interval); unit: mL/kg/min
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 10 | 10
mL/kg/min | 3.5 [1.2 to 5.9] | 1.7 [0.03 to 3.3]

5. Secondary Outcome: Change in VE/VCO2 From Baseline to Week 12
Description: VE/VCO2 is assessed from cardiopulmonary exercise testing results.
Time Frame: Baseline and Week 12
Measure: Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 10 | 10
Ratio | -2.2 [-6.1 to 1.7] | -2.5 [-4.3 to -0.7]

6. Secondary Outcome: Change in Resting LVEF From Baseline to Week 12
Description: LVEF is assessed by echocardiography.
Time Frame: Baseline and Week 12
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 10 | 10
Percent change | -14.6 [-23.1 to -6.2] | -5.5 [-9.8 to -1.2]

7. Secondary Outcome: Change in LV Fractional Shortening (LVFS) From Baseline to Week 12
Description: LVFS is assessed using echocardiography measures.
Time Frame: Baseline and Week 12
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 10 | 8
Percent | -18.60 (13.05) | -3.98 (11.42)

8. Secondary Outcome: Change in Global Longitudinal Strain (GLS) From Baseline to Week 12
Description: GLS is assessed using echocardiography measures.
Time Frame: Baseline and Week 12
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 9 | 10
Percent | 0.56 (3.778) | 0.18 (2.806)

9. Secondary Outcome: Change in Post-exercise Peak LVOT Gradient From Week 12 to Week 16
Description: Post-exercise peak LVOT gradients are assessed after a treadmill stress test by echocardiography.
Time Frame: Weeks 12 and 16
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 8 | 10
mm Hg | 55.22 (40.84) | 84.08 (28.38)

10. Other Pre Specified Outcome: Change in NYHA Functional Class From Baseline to Week 12
Time Frame: Baseline and Week 12
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Change in KCCQ OSS From Baseline to Week 12
Time Frame: Baseline and Week 12
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Change in NT-proBNP From Baseline to Week 12
Time Frame: 12 weeks
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Number of Subjects Achieving an LVOT Gradient Response of Post-exercise Peak Gradient < 10 mmHg at Week 12
Description: Post-exercise peak LVOT gradients are assessed after a treadmill stress test by echocardiography.
Time Frame: Baseline and Week 12
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 16 Weeks
Description: Adverse event data were collected from baseline through the end of study visit at Week 16 for each participant enrolled.
Arm/Group | Cohort A | Cohort B
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/11 | 0/10
Other Adverse Events (participants affected / at risk) | 10/11 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=11) | Cohort B (N=10)
Atrial Fibrillation (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=11) | Cohort B (N=10)
Ventricular Tachycardia (Cardiac disorders) | 1 | 4
Atrial Fibrillation (Cardiac disorders) | 3 | 1
Headache (Nervous system disorders) | 3 | 2
Dizziness (Nervous system disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 2 | 0
Angina Pectoris (Cardiac disorders) | 0 | 2
Fatigue (General disorders) | 2 | 2
Application Site Rash (General disorders) | 0 | 2
Dyspnea (Exertional) (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 2
Urinary Tract Infection (Infections and infestations) | 2 | 0
Ejection Fraction Decreased (Investigations) | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Cardiac Failure (Cardiac disorders) | 1 | 0
Cardiac Flutter (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Food Poisoning (Gastrointestinal disorders) | 1 | 0
Gastric Ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Retching (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1
Application Site Erythema (General disorders) | 1 | 0
Asthenia (General disorders) | 1 | 1
Chills (General disorders) | 1 | 0
Feeling Abnormal (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Peripheral Swelling (General disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Heat exhaustion (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Blood calcium decreased (Investigations) | 0 | 1
Blood creatine phosphokinase abnormal (Investigations) | 1 | 0
Brain natriuretic peptide increased (Investigations) | 1 | 1
Heart rate irregular (Investigations) | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Hypersomnia (Nervous system disorders) | 0 | 1
Hyporeflexia (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Breast mass (Reproductive system and breast disorders) | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's have the right to publish data after the primary publication is released.

DOCUMENTS (2):
  • Study Protocol (2017-05-05): https://cdn.clinicaltrials.gov/large-docs/42/NCT02842242/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-24): https://cdn.clinicaltrials.gov/large-docs/42/NCT02842242/SAP_001.pdf